CLINICAL TRIAL: NCT00938002
Title: Rapid Bacterial Identification and Antibiotic Resistance Testing in Critically Ill Adults at Risk for Ventilator Acquired Pneumonia (VAP).
Brief Title: Study to Determine Quicker Methods of Diagnosing Pneumonia Caused by a Breathing Machine in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: Accerl8 Technology Corporation (Other); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Ivor Douglas, Chief, Pulmonary Sciences & Critical Care Medicine, Denver Health and Hospital Authority
Other Study IDs: 09-0321; UL1RR025780 (NIH)
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Ventilator Acquired Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA collected from whole blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Diagnostic Test: Acceler8 Pheno

SUMMARY:
Critically ill patients on a breathing machine are at risk of developing a type of pneumonia called Ventilator Acquired Pneumonia (VAP). The purpose of this study is to determine if regular lung rinses sent for microbiological testing can reduce the time to diagnose VAP. The study also plans to test the accuracy and speed of a new technology, using multiplexed automated digital microscopy, to identify the germs causing the VAP.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP) is a common, life-threatening hospital-acquired infectious complication of prolonged mechanical ventilation (MV). Despite aggressive efforts to prevent VAP, rates remain high because clinical diagnosis is imprecise and microbiological diagnosis is frequently delayed. Diagnosis of VAP depends on clinical signs as well as microbiologic evidence from Bronchioalveolar Lavage (BAL) cultures. Ordinarily, these cultures are only ordered after the patient presents with clinical signs and symptoms of VAP, which can significantly delay diagnosis and effective therapy. This research proposes to implement additional surveillance BAL cultures in order to reduce the time to diagnosis of VAP in mechanically ventilated critically ill adults. To further reduce the time to diagnosis of VAP, this research aims to test part of the BAL cultures using a novel flowcell/surface-capture device that allows direct from specimen visualization of bacteria using multiplexed automated digital microscopy (BACcel™) for rapid bacterial identification and antibiotic resistance testing. Additionally, molecular assays of the BAL sample will characterize lower respiratory tract antimicrobial peptide host-innate immune molecule and local anti-oxidant defenses in mechanically ventilated adults at risk for VAP.

ELIGIBILITY:
Inclusion Criteria:

1. Written, informed consent (by surrogate if unconscious or if altered mental status)
2. ≥ 18 years old
3. Admission to a Medical Intensive care unit
4. Orally/nasally intubated, evaluable within 72 h of initial intubation
5. Expected to remain mechanically ventilated for at least 48 h after the first study procedure

Exclusion Criteria:

1. Previously documented cystic fibrosis
2. Diffuse bronchiectasis
3. Severe or massive hemoptysis
4. Presence of an advanced directive to withhold life-sustaining treatment
5. Morbid state or expected to survive less than 14 days because of an advanced co-morbid medical condition
6. Participation in a clinical trial of any unlicensed drug or device within 30 days
7. Pregnant or Nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill ventilated patients
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2009-07; Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Reduction in time to diagnosis and treatment of VAP in an at risk population | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Ivor S Douglas, MD, Principal Investigator — Denver Health and Hospital Authority; Connie S Price, MD, Principal Investigator — Denver Health and Hospital Authority
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No